CLINICAL TRIAL: NCT00189540
Title: A Phase II Double-Blind, Randomized, Placebo-Controlled Study to Assess the Safety and Efficacy of AMG0001 to Improve Perfusion in Critical Limb Ischemia in Subjects Who Have Peripheral Ischemic Ulcers
Brief Title: Study of Hepatocyte Growth Factor (HGF) Via Plasmid Vector to Improve Perfusion in Critical Limb Ischemia Patients With Peripheral Ischemic Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AnGes USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG-CLI-0205
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Arterial Occlusive Disease; Peripheral Vascular Disease; Ischemia; Ulcers
Keywords: Ischemic ulcers; Critical Limb Ischemia
MeSH Terms: conditions — Arterial Occlusive Diseases; Peripheral Vascular Diseases; Ischemia; Ulcer; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Active Group (Active Comparator): 4.0 mg AMG0001 via intramuscular injections on days 0, 14, and 28
  Interventions: Genetic: HGF plasmid
- Placebo Group (Placebo Comparator): Placebo (saline) via intramuscular injections on days 0, 14, and 28
  Interventions: Genetic: Placebo

INTERVENTIONS:
Genetic: HGF plasmid — Intramuscular injections into the index leg on days 0, 14, and 28
  Arms: Active Group
Genetic: Placebo — Intramuscular injections into the index leg on days 0, 14, and 28
  Arms: Placebo Group

SUMMARY:
The objective of this study is to test the hypothesis that AMG0001 treatment is safe and induces angiogenesis as detected by improved wound healing, reduction in amputation, improved pain at rest and hemodynamic measurement and to assess the effectiveness of the administrative method.

DETAILED DESCRIPTION:
The primary goals of this study evaluating AMG0001 administration in CLI subjects will be to investigate the efficacy and safety of AMG0001. Specifically, the objectives are:

1. Assess efficacy of a dosing regimen of 4.0mg/3 mL AMG0001, administered on Days 0, 14, and 28 as measured by reduction in total wound area at Month 3.
2. Assess potential effects of angiogenesis associated with a dosing regimen of 4.0mg/3 mL AMG0001, administered on Days 0, 14, and 28 as measured by reduction in total wound area at Months 6 and 12, along with reduction in major amputations and improved pain at rest as measured on the VAS and hemodynamic measures (ABI/TBI) at Month 3 and Month 6.
3. Assess overall safety of AMG0001 in the Critical Limb Ischemia subject population as determined by physical examination, blood and urine analyses, electrocardiogram, vital signs, and by evaluation of adverse experiences during and after the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will have an appropriately sized peripheral ischemic ulcer(s).
2. Subjects will have one or both of the following hemodynamic indicators of severe peripheral arterial occlusive disease:

   1. Ankle systolic pressure (in either the dorsalis pedis or posterior tibial arteries) of < 70 mmHg
   2. Toe systolic pressure < 50 mmHg
3. The subject is a poor candidate for standard revascularization treatment options for peripheral arterial disease, based on inadequate bypass conduit, unfavorable anatomy, or poor operative risk.
4. Subjects 40 years or older of either sex who have signed an informed consent form either directly or through a legally authorized representative.
5. Subjects will be on a statin and an anti-platelet agent (e.g., clopidogrel, ticlopidine, aspirin, etc.) as part of their standard of care, unless contraindicated. Subjects for which these agents are contraindicated will have this restriction recorded in their case report form (CRF). Subjects must be stable on these medical regimens for at least 4 weeks prior to the start of treatment.
6. If female, the subjects must be:

   1. at least one year post-menopausal, or
   2. surgically sterile, or
   3. if the subject is of child-bearing potential, she must have been practicing adequate contraception for at least 12 weeks prior to entering the study and have a negative urine pregnancy test result prior to study enrollment and agree to periodic pregnancy screening tests during the study.
   4. If female, the subject must not be breastfeeding for 30 days following administration of HGF.
7. If subject is of reproductive potential, he or she must be using an accepted and effective (barrier) form of birth control during the study.

Exclusion Criteria

1. Subjects who, in the opinion of the investigator, have a vascular disease prognosis that indicates they would require a major amputation (at or above the ankle) within 4 weeks of start of treatment.
2. Subjects with a diagnosis of Buerger's disease (thromboangiitis obliterans).
3. Subjects with hemodynamically significant aorto-iliac occlusive disease.
4. Subjects who have had a revascularization procedure within 12 weeks prior to treatment initiation that remains patent. Revascularization procedures that are evidenced to have failed (completely occluded) for >2 weeks prior to treatment initiation are acceptable.
5. Subjects who require a change in their hypertension medication (other than dosage change) as part of their standard of care within 4 weeks prior to treatment initiation.
6. Subjects with deep ulcerations with bone or tendon exposure, or clinical evidence of invasive infection (e.g., cellulitis, osteomyelitis, etc.) uncontrollable by antibiotics.
7. Subjects currently receiving immuno-suppressive medication, chemo or radiation therapy.
8. Evidence or history of malignant neoplasm (clinical, laboratory or imaging), except for fully resolved basal cell carcinoma of the skin. Patient's who had successful tumor resection or radio-chemotherapy of breast cancer more than 10 years prior to inclusion in the study, and with no recurrence, may be enrolled in the study. Patient's who had successful tumor resection or radio-chemotherapy of all other tumor types more than 5 years prior to inclusion in the study, and with no recurrence, may be enrolled in the study.
9. Subjects who have proliferative diabetic retinopathy, severe non-proliferative retinopathy, recent (within 6 months) retinal vein occlusion, macular degeneration with choroidal neovascularization, macular edema on fundus evaluation by ophthalmologist, or intraocular surgery within 3 months.
10. Subjects with end stage renal disease (ESRD) defined as significant renal dysfunction evidenced by a creatinine of > 2.5 mg/dL, or receiving chronic hemodialysis therapy.
11. Any co-morbid condition likely to interfere with assessment of safety or efficacy endpoints, acute cardiovascular events (i.e. cerebrovascular accident [CVA], myocardial infarction [MI], etc.) within 12 weeks of treatment, or non-cardiovascular diseases that in the opinion of the investigator may result in < 3 month subject mortality.
12. A subject who has a history of hepatic cirrhosis, viral hepatitis, or HIV.
13. Subjects with a clinically significant liver enzyme abnormality (i.e., AST or ALT more than two times the upper limit of normal and/or bilirubin more than 50% above the upper limit of normal).
14. Subjects taking cilostazol (Pletal®) are eligible for inclusion, but the subject must have been taking the medication for at least 4 weeks prior to test material administration.
15. Subject who received another investigational drug for peripheral arterial disease within 90 days of randomization, have previously received any gene transfer therapy or growth factor product not approved by the United States Food and Drug Administration (FDA) or received any investigational Drug Product in another clinical trial in the 30 days prior to administration of HGF.
16. Unreliable or uncooperative subject or other severe concomitant disease(s), which the clinical investigator feels constitute(s) criteria for exclusion of a particular subject.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-08; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Powell, MD, Principal Investigator — Dartmouth
Locations (4):
- United States (4):
  - Baptist Clinical Research, Pensacola, Florida
  - The Care Group, LLC, Indianapolis, Indiana
  - Boston Medical Center, Boston, Massachusetts
  - Dartmouth - Hitchcock Medical Center, Lebanon, New Hampshire

REFERENCES:
- [Result] Powell RJ, Goodney P, Mendelsohn FO, Moen EK, Annex BH; HGF-0205 Trial Investigators. Safety and efficacy of patient specific intramuscular injection of HGF plasmid gene therapy on limb perfusion and wound healing in patients with ischemic lower extremity ulceration: results of the HGF-0205 trial. J Vasc Surg. 2010 Dec;52(6):1525-30. doi: 10.1016/j.jvs.2010.07.044. PMID 21146749

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening was up to 30 days
Groups:
- Active Group: 4.0 mg AMG0001 via IM injections on days 0, 14, and 28
- Placebo Group: Placebo (saline)via IM injections on days 0, 14, and 28
Period: Overall Study
Arm/Group | Active Group | Placebo Group
Started | 21 | 6
Completed | 14 | 5
Not Completed | 7 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Death | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Group | Placebo Group | Total
Number analyzed (Participants) | 21 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.7 (2.49) | 78.0 (1.86) | 76.2 (1.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 13 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Wound Healing (Change in Total Wound Area of All Ischemic Ulcers)
Description: Wound healing measured by change in mean total wound area of all ischemic ulcers at Month 3 and Month 6
Time Frame: Baseline, Month 3, Month 6
Population: Per protocol population - Efficacy Evaluable or EE
Measure: Mean (Standard Error); unit: total wound area (cm^2)
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 16 | 5
total wound area (cm^2)
  Baseline | 5.75 (1.8134) | 12.600 (9.4435)
  Month 3 | 15.766 (6.8421) | 12.200 (8.7022)
  Month 6 | 16.375 (7.1336) | 12.700 (9.7190)
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Comparison made is the difference from baseline at Month 3; Test type: Superiority or Other; p = 0.35, ANCOVA
Statistical Analysis 2: Comparison: Active Group vs Placebo Group; Comparison made is the difference from baseline at Month 6; Test type: Superiority or Other; p = 0.17, ANCOVA

2. Secondary Outcome: Percentage of Participants Where All Ulcers Healed
Description: This outcome is a percentage of participants where all of their baseline ulcers healed.
Time Frame: Month 3 and Month 6
Population: Per protocol population Efficacy Evaluable "EE"
Measure: Number; unit: Percentage of Participants
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 16 | 5
Percentage of Participants
  Month 3 | 6 | 0
  Month 6 | 19 | 0
  Month 12 | 31 | 0
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; The comparison of groups at Month 3; Test type: Superiority or Other; p = 0.55, Fisher Exact
Statistical Analysis 2: Comparison: Active Group vs Placebo Group; The comparison of groups at Month 6; Test type: Superiority or Other; p = 0.28, Fisher Exact

3. Secondary Outcome: Change in Pain at Rest as Measured on the Visual Analog Scale (VAS)
Description: The mean VAS score where 0 = no pain; 10 = worst possible pain.
Time Frame: Baseline, Month 3 and Month 6
Population: Per protocol population or Efficacy Evaluable "EE"
Measure: Mean (Standard Error); unit: cm
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 16 | 5
cm
  Baseline | 5.31 (0.60) | 6.04 (1.20)
  Month 3 | 4.26 (0.92) | 6.52 (1.5)
  Month 6 | 3.40 (0.99) | 6.66 (1.3)
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Comparison between groups at Month 3; Test type: Superiority or Other; p = 0.2, ANCOVA
Statistical Analysis 2: Comparison: Active Group vs Placebo Group; Comparison between groups at Month 6; Test type: Superiority or Other; p = 0.04, ANCOVA

4. Secondary Outcome: Number of Subjects Who Undergo a Major Amputation
Time Frame: Month 3 and Month 6
Measure: Number; unit: participants
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 16 | 5
participants
  3 months | 3 | 0
  6 months | 3 | 0
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Test type: Superiority or Other; p = 1.00, Fisher Exact

5. Secondary Outcome: Change in Hemodynamic Measurements - Mean Change in Ankle Brachial Index (ABI)
Time Frame: Baseline, Month 3, Month 6
Population: Population is per protocol - Efficacy Evaluable (EE)
Measure: Mean (Standard Error); unit: mm Hg / mm Hg
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 16 | 5
mm Hg / mm Hg
  Baseline | 0.492 (0.0662) | 0.430 (0.0957)
  Month 3 | 0.476 (0.0657) | 0.448 (0.1248)
  Month 6 | 0.472 (0.0846) | 0.303 (0.1481)
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Comparison at Month 3; Test type: Superiority or Other; p = 0.77, ANCOVA
Statistical Analysis 2: Comparison: Active Group vs Placebo Group; Comparison at Month 6; Test type: Superiority or Other; p = 0.45, ANCOVA

6. Secondary Outcome: Change in Hemodynamic Measurements - Mean Change in Toe Brachial Index (TBI)
Time Frame: Baseline, Month 3, Month 6
Population: Population is per protocol - Efficacy Evaluable (EE)
Measure: Mean (Standard Error); unit: mm Hg / mm Hg
Arm/Group | Active Group | Placebo Group
Number analyzed (Participants) | 16 | 5
mm Hg / mm Hg
  Baseline | 0.19 (0.04) | 0.28 (0.06)
  Month 3 | 0.22 (0.05) | 0.14 (0.06)
  Month 6 | 0.24 (0.06) | 0.11 (0.07)
Statistical Analysis 1: Comparison: Active Group vs Placebo Group; Comparison between groups for mean TBI at Month 3 versus baseline; Test type: Superiority or Other; p = 0.06, ANCOVA
Statistical Analysis 2: Comparison: Active Group vs Placebo Group; Comparison between groups for mean TBI at Month 6 versus baseline; Test type: Superiority or Other; p = 0.05, ANCOVA

ADVERSE EVENTS:
Arm/Group | Active Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 17/21 | 3/6
Other Adverse Events (participants affected / at risk) | 20/21 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Group (N=21) | Placebo Group (N=6)
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Death (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Lobar Pneumonia (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Mental Status Change (Psychiatric disorders) | 1 | 0
Knee Arthroplasty (Surgical and medical procedures) | 1 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0
Ischaemic ulcer (Vascular disorders) | 1 | 0
Peripheral Arterial occlusive disease (Vascular disorders) | 9 | 2
Localised Infection (Infections and infestations) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Group (N=21) | Placebo Group (N=6)
Anaemia (Blood and lymphatic system disorders) | 7 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 1
Injection Site Discomfort (General disorders) | 2 | 0
Oedema Peripheral (General disorders) | 5 | 1
Pyrexia (General disorders) | 5 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 3
Localised infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 5 | 0
Sepsis (Infections and infestations) | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 4 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 1 | 1
Blood uric acid increased (Investigations) | 0 | 1
Chest x-ray abnormal (Investigations) | 2 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 1
Electrocardiogram abnormal (Investigations) | 2 | 1
International normalised ratio increased (Investigations) | 2 | 0
Occult blood positive (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 2
Depressed level of conciousness (Nervous system disorders) | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 2 | 0
Auditory hallucination (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 0
Renal impairment (Renal and urinary disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 1
Ischaemic limb pain (Vascular disorders) | 2 | 0
Ischaemic ulcer (Vascular disorders) | 8 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 11 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Multi-center all inclusive initial publication planned. Any proposed publications must be submitted to the steering committee and sponsor thirty (30) days prior to publication submission.